CLINICAL TRIAL: NCT00710242
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Assess the Safety and Efficacy or Pre-Treatment With DF01 During Late Pregnancy in Reducing Prolonged Labor
Brief Title: Study to Assess Safety and Efficacy of DF01 in Reducing Prolonged Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dilafor AB (Industry)
Responsible Party: Clinical Research Director, Dilafor AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPL02
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Pregnancy; Labor
Keywords: prolonged labor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DF01
  Interventions: Drug: DF01
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DF01 — Once daily s.c. injections from approximately 3-7 days before expected delivery (maximum 2 weeks before) until delivery (maximum 2 weeks after expected delivery)
  Arms: 1
Drug: Placebo — Once daily s.c. injections from approximately 3-7 days before expected delivery (maximum 2 weeks before) until delivery (maximum 2 weeks after expected delivery)
  Arms: 2

SUMMARY:
The study is a Proof-of-concept study to evaluate if DF01 can prevent protracted labor. Time to delivery will be measured from the time of at least 3 cm cervix dilatation and 3 contractions of minimum one minute's duration/10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy nulliparous females
* normal singleton pregnancy
* intact membranes

Exclusion Criteria:

* breech or other abnormal presentation
* intercurrent illness
* pregnancy complications
* vaginal bleeding in third trimester
* etc

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Time from the time of at least 3 cm cervix dilatation and 3 contractions of minimum one minute's duration/10 minutes until partus in women with vaginal delivery | See above

SECONDARY OUTCOMES:
Complications of labor | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lena Granstrom, MD, Principal Investigator — Kvinnokliniken Sodra Alvsborgs sjukhus Boras; Gunvor Ekman-Ordeberg, MD, PhD, Study Chair — Dilafor AB
Locations (18):
- Sweden (18):
  - Kvinnokliniken Alvsborgs sjukhus Boras, Borås
  - Gavle sjukhus, Gävle
  - Sahlgrenska/Ostra sjukhuset, Gothenburg
  - Karolinska Universistetssjuhuset, Huddinge
  - Lanssjukhuset Ryhov, Jönköping
  - Lanssjukhuset, Kalmar
  - Universitetssjukhuset, Linköping
  - Universitetssjukhuset, Lund
  - Vrinnevisjukhuset, Norrköping
  - Nyköpings lasarett, Nyköping
  - Universitetssjukhuset, Örebro
  - Kärnsjukhuset, Skövde
  - Danderyds sjukhus, Stockholm
  - Sodersjukhuset, Stockholm
  - Norra Älvsborgs länssjukhus, Trollhättan
  - Akademiska sjukhuset, Uppsala
  - Centrallasarettet, Vaxjo
  - Centrallasarettet, Västerås

REFERENCES:
- [Derived] Ekman-Ordeberg G, Hellgren-Wangdahl M, Jeppson A, Rahkonen L, Blomberg M, Pettersson K, Bejlum C, Engberg M, Ludvigsen M, Uotila J, Tihtonen K, Hallberg G, Jonsson M. Tafoxiparin, a novel drug candidate for cervical ripening and labor augmentation: results from 2 randomized, placebo-controlled studies. Am J Obstet Gynecol. 2024 Mar;230(3S):S759-S768. doi: 10.1016/j.ajog.2022.10.013. Epub 2023 May 17. PMID 38462256